CLINICAL TRIAL: NCT03039127
Title: Interstitial Laser Thermotherapy (imILT) as a Treatment Option in Breast Cancer Patients Not Suitable for Surgical Excision
Brief Title: Immunostimulating Interstitial Laser Thermotherapy in Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped in agreement with investigator due to slow recruitment.
Sponsor: Clinical Laserthermia Systems AB (Industry)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-2015-009
Record Dates: First submitted 2016-06-29; First posted 2017-02-01 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Breast Neoplasms
Keywords: Hyperthermia; Laser Coagulation; Laser Therapy; Induced
MeSH Terms: conditions — Breast Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imILT (Experimental): Immunostimulating Interstitial Laser Thermotherapy (imILT)
  Interventions: Device: Immunostimulating Interstitial Laser Thermotherapy

INTERVENTIONS:
Device: Immunostimulating Interstitial Laser Thermotherapy — Immunostimulating Interstitial Laser Thermotherapy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response.

SUMMARY:
Thermotherapy is a technology aiming at destroying tissue, for example tumor tissue. Immunostimulating Interstitial Laser Thermotherapy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response. In laboratory animals the imILT method has also been shown to induce a so called abscopal effect. This means that when one tumor is treated with imILT other, untreated, tumors also decrease in size. The immunologic response has previously been characterized in breast cancer patients after receiving imILT treatment , and presumed abscopal effects induced by imILT have also been described in a malignant melanoma patient.

The purpose of this trial is to investigate the functionality and safety of the imILT treatment method in patients diagnosed with breast cancer.

The treatment method has successfully been used for treatment of patients with breast cancer and malignant melanoma. Treatment of breast cancer patients caused an increase of cytotoxic T lymphocytes in the treated tumor, as well as activated dendritic cells at the tumor border. Regulatory T lymphocytes decreased in the regional lymph nodes.

This trial is explorative, prospective, open and non-randomized. Five breast cancer patients will be treated in this trial, which is estimated to be carried out during a time period of 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed breast cancer
2. Hormone receptor positive or negative
3. Have assessable tumour by MRI or ultrasound
4. Are patients deemed unfit for surgical excision of tumour under general anaesthetic.
5. Have been given informed verbal and written consent for participation in the trial
6. Have stable hematologic, renal and hepatic functions.

Exclusion Criteria:

1. Are known to be HIV positive
2. Have active autoimmune disease
3. Are on corticosteroid medication
4. Have evidence of bleeding diathesis or coagulopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-06; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Treatment effect by radiology | 9 months
  Evaluation by Response Evaluation Criteria in Solid Tumours (RECIST)

SECONDARY OUTCOMES:
Safety (adverse events) | 9 months
  Evaluation of adverse events and laboratory analyses.
Usability (user evaluation of instrument) | 9 months
  Analysis of instrument and user questionnaires relating to the ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: Kristjan S Asgeirsson, MD, Principal Investigator — Nottingham Breast Institute
Locations (1):
- Nottingham Breast Cancer Institute, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haraldsdottir KH, Ingvar C, Stenram U, Tranberg KG. Long-term Follow-up After Interstitial Laser Thermotherapy of Breast Cancer. Anticancer Res. 2015 Nov;35(11):6147-52. PMID 26504041
- [Result] Haraldsdottir KH, Ivarsson K, Jansner K, Stenram U, Tranberg KG. Changes in immunocompetent cells after interstitial laser thermotherapy of breast cancer. Cancer Immunol Immunother. 2011 Jun;60(6):847-56. doi: 10.1007/s00262-011-0992-8. Epub 2011 Mar 13. PMID 21400025
- [Result] Ivarsson K, Myllymaki L, Jansner K, Stenram U, Tranberg KG. Resistance to tumour challenge after tumour laser thermotherapy is associated with a cellular immune response. Br J Cancer. 2005 Aug 22;93(4):435-40. doi: 10.1038/sj.bjc.6602718. PMID 16091763
- [Result] Tranberg KG, Moller PH, Hannesson P, Stenram U. Interstitial laser treatment of malignant tumours: initial experience. Eur J Surg Oncol. 1996 Feb;22(1):47-54. doi: 10.1016/s0748-7983(96)91451-1. PMID 8846867
- [Result] Tranberg KG, Myllymaki L, Moller PH, Ivarsson K, Sjogren HO, Stenram U. Interstitial laser thermotherapy of a rat liver adenocarcinoma. J Xray Sci Technol. 2002 Jan 1;10(3):177-85. PMID 22388047
- [Result] Ivarsson K, Myllymaki L, Jansner K, Bruun A, Stenram U, Tranberg KG. Heat shock protein 70 (HSP70) after laser thermotherapy of an adenocarcinoma transplanted into rat liver. Anticancer Res. 2003 Sep-Oct;23(5A):3703-12. PMID 14666667